CLINICAL TRIAL: NCT04217096
Title: A Single-arm, Prospective Study to Evaluate the Efficacy and Safety of the Combination of Paclitaxel Liposome and S-1 as First-line Therapy in Treating Patients With Advanced Metastatic Pancreatic Cancer
Brief Title: Efficacy and Safety of Paclitaxel Liposome and S-1 as First-line Therapy in \ Advanced Pancreatic Cancer Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, Principal Investigator, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPAC-21
Record Dates: First submitted 2019-12-31; First posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Advanced Pancreatic Cancer
MeSH Terms: interventions — S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- paclitaxel liposome + S-1 (Experimental): paclitaxel liposome at 175 mg/m^2 on day 1; S-1 at a dose according to the body surface area（<1.25m^2，40mg Bid；1.25~1.5m^2,50mg Bid；>1.50m^2,60mg Bid，d1-14，q3w）
  Interventions: Drug: Paclitaxel liposome; Drug: S-1

INTERVENTIONS:
Drug: Paclitaxel liposome — Patients receive paclitaxel liposome 175 mg/m^2 (iv, 3h) on day 1 for 3 weeks. Treatment repeats every 3 weeks until the disease recurrence or unacceptable toxicity，death or begin a novel therapeutic
Drug: S-1 — Patients receive S-1 at a dose according to the body surface area（<1.25m^2，40mg Bid；1.25~1.5m^2,50mg Bid；>1.50m^2,60mg Bid）on days 1-14 for 3 weeks. Treatment repeats every 3 weeks until the disease recurrence or unacceptable toxicity，death or begin a novel therapeutic.

SUMMARY:
The present study is intended to investigate the efficacy and safety of the patients with confirmed advanced pancreatic cancer after treating with the combination of paclitaxel liposome plus S-1.

DETAILED DESCRIPTION:
Allocation: Non-randomized Endpoint Classification: Efficacy/ Safety Study Intervention Model: single arm Masking: Open Lable Primary Purpose: Treatment

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤75 years;
2. the patients were confirmed as locally advanced or metastatic pancreatic cancer by histopathology;
3. At least one measurable objective lesion was identified based on the RECIST1.1 criteria;
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
5. The expected survival after surgery ≥3 months;
6. Adequate liver/kidney/bone marrow function： Absolute neutrophil count (ANC) ≥1.5×10^9/L; Hemoglobin (Hgb) ≥9g/dL; Platelets (PLT) ≥100×10^9/L; Total bilirubin (TBIL) ≤1.5×ULN; Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]/ alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) ≤2.5×institutional upper limit of normal (ULN), or ≤5×ULN(hepatic metastases); Serum creatinine level is normal or creatinine clearance rate≥60 mL/min/1.73 m^2.
7. Subjects of child-bearing age must agree to take effective contraceptive measures during the study period; Serum or urine pregnancy tests must be negative for women of childbearing age 7 days before the start of chemotherapy、during the monthly treatment interval and after the last treatment;
8. Signed informed content obtained prior to treatment.

Exclusion Criteria:

1. Symptomatic ascites;
2. The target disease has cerebral metastasis;
3. Previously received palliative chemotherapy or other palliative systemic therapy for advanced/metastatic pancreatic cancer;
4. Previously received treatments based on paclitaxel liposomes or S-1, except for neoadjuvant therapy or adjuvant therapy (before and after R0/R1 excision), which was based on paclitaxel liposomes or S-1(the time of discontinuation of neoadjuvant/adjuvant chemotherapy before admission ≥6 months);
5. Received surgical treatment ≤4 weeks before admission;
6. Severe cancer-related cachexia and/or known weight loss >15% occurred within one month before admission;
7. The medical history and complications, which may affect patients' ability to participate in the study and their safety during the study, or interfere with explanation of the study results, for example: uncontrolled hypertension, cardiovascular and cerebrovascular diseases such as cerebrovascular accident (≤6 months from the start of the study), myocardial infarction (≤less than 6 months from the start of the study), unstable angina pectoris, heart failure (≥2 grades) (NYHA functional score), severe arrhythmia requiring medication, metabolic dysfunction, severe renal insufficiency;
8. Human immunodeficiency virus (HIV) or Hepatitis B Virus（HBV）、hepatitis C virus (HCV) positive with Liver dysfunction;
9. Combined with other malignant tumors excepted pancreatic cancer within the first 5 years of admission, excepted cured carcinoma in situ of cervix、basal cell carcinoma of the skin;
10. History of allergy or hypersensitivity to any therapeutic ingredient;
11. Patients with known active alcohol or drug abuse or dependence;
12. Pregnancy, or women who are currently trying to conceive, or who are likely to have children and do not use contraceptives, or breastfeeding women;
13. Participation in any trial drug treatment or another interventional clinical trial 30 days before screening period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | from the date of enrollment to the day of progression or death of any cause, whichever come first, assessed up to 10 months
  To evaluate the Progression Free Survival of patients with advanced pancreatic cancer after treated with paclitaxel liposome plus S-1.

SECONDARY OUTCOMES:
Overall Response Rate | from the date of enrollment to the day of progression or death of any cause, whichever come first, assessed up to 10 months
  To evaluate the Overall Response Rate of patients with advanced pancreatic cancer after treated with paclitaxel liposome plus S-1.
overall survival | from the date of enrollmen to death of any cause or the end of this trial, whichever come first, assessed up to 10 months
  To evaluate the overall survival of patients with advanced pancreatic cancer after treated with paclitaxel liposome plus S-1.
Disease control rate | from the date of enrollment to the day of progression or death of any cause, whichever come first, assessed up to 10 months
  To evaluate the disease control rate of patients with advanced pancreatic cancer after treated with paclitaxel liposome plus S-1.
Quality of life (Qol) | from the date of enrollmen to death of any cause or the end of this trial, whichever come first, assessed up to 10 months
  To evaluate the Quality of Life of patients with advanced pancreatic cancer after treated with paclitaxel liposome plus S-1.
Adverse events | from the date of enrollmen to death of any cause or the end of this trial, whichever come first, assessed up to 10 months
  To evaluate the adverse events of patients with advanced pancreatic cancer after treated with paclitaxel liposome plus S-1.

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Jun Yu, M.D., Ph.D., Principal Investigator — Fudan University
Locations (1):
- Department of Pancreatic and Hepatobiliary Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University; 270 Dong An Road, Shanghai 200032, China, Shanghai, China

IPD SHARING:
Plan to Share IPD: No